CLINICAL TRIAL: NCT01535261
Title: A 24-month, Phase IIIb, Open-label, Single Arm, Multicenter Study Assessing the Efficacy and Safety of an Individualized, Stabilization-criteria-driven PRN Dosing Regimen With 0.5-mg Ranibizumab Intravitreal Injections Applied as Monotherapy in Patients With Visual Impairment Due to Macular Edema Secondary to Central Retinal
Brief Title: Ranibizumab Intravitreal Injections in Patients With Visual Impairment Due to Macular Edema Secondary to Central Retinal Vein Occlusion
Acronym: CRYSTAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002E2401; 2011-002350-31 (EudraCT Number)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Macular Edema; Central Retinal Vein Occlusion
Keywords: Ophthalmology; Ranibizumab; Central Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab

ARMS (1):
- Ranibizumab arm (Experimental): Intravitreal injection with standard dose of 0.5 mg/0.05mL PRN
  Interventions: Drug: Ranibizumab 0.5 mg/0.05 ml

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg/0.05 ml — Patients will receive the first dose at Baseline, as an intravitreal injection with a standard dose of 0.5 mg/0.05 ml. Patients will receive at least 3 study treatments at monthly intervals (Day 1, Month 1 and Month 2). The last mandatory dose during treatment initiation will be administered approximately 60 days after the first study treatment. If there is no improvement in VA over the course of the first 3 injections, continued treatment is not recommended and the patient may receive alternative treatment at the investigator's discretion.

SUMMARY:
The present study provided additional efficacy and safety data for 0.5-mg ranibizumab using as needed (PRN) dosing over 24 months in patients with visual impairment due to macular edema secondary to Central Retinal Vein Occlusion (CRVO). Spectral domain high-definition optical coherence tomography (OCT) images was analyzed to gain insights into predictive factors for disease progression and the possibility of reduced monitoring was assessed in Year 2. The results of this open-label study provided long-term safety and efficacy data to further guide recommendations on the use of ranibizumab in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age
* Diagnosis of visual impairment exclusively due to ME secondary to CRVO
* BCVA score at Screening and Baseline between 73 and 19 letters Early Treatment Diabetic Retinopathy Study (ETDRS), inclusively (approximate Snellen chart equivalent of 20/40 and 20/400)

Exclusion Criteria:

* Uncontrolled blood pressure defined as systolic value of > 160 mm Hg or diastolic value of > 100 mm Hg at Screening or Baseline.
* Any active periocular or ocular infection or inflammation at Screening or Baseline in either eye
* Uncontrolled glaucoma at Screening or Baseline or diagnosed within 6 months before Baseline in either eye
* Use of any systemic antivascular endothelial growth factor (anti-VEGF) drugs within 6 months before Baseline (eg, sorafenib [Nexavar®], sunitinib [Sutent®], bevacizumab [Avastin®])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- Australia (4):
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Vienna, Austria
  - Novartis Investigative Site, Linz
- Canada (6):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Glostrup Municipality, Denmark
- Greece (6):
  - Novartis Investigative Site, Pátrai, Greece
  - Novartis Investigative Site, Thessaloniki, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion Crete, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Ireland (2):
  - Novartis Investigative Site, Dublin, Ireland
  - Novartis Investigative Site, Dublin
- Italy (6):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine
- Netherlands (5):
  - Novartis Investigative Site, Leiden 2333 ZA, Netherlands
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Tilburg
- Poland (6):
  - Novartis Investigative Site, Bielsko-Biala
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (4):
  - Novartis Investigative Site, Porto, Porto District
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Lisbon
- Slovakia (3):
  - Novartis Investigative Site, Žilina, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Banská Bystrica
- Spain (7):
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Örebro, Sweden
- Switzerland (3):
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
- Novartis Investigative Site, Ankara, Turkey, Turkey (Türkiye)
- United Kingdom (11):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Pawloff M, Bogunovic H, Gruber A, Michl M, Riedl S, Schmidt-Erfurth U. SYSTEMATIC CORRELATION OF CENTRAL SUBFIELD THICKNESS WITH RETINAL FLUID VOLUMES QUANTIFIED BY DEEP LEARNING IN THE MAJOR EXUDATIVE MACULAR DISEASES. Retina. 2022 May 1;42(5):831-841. doi: 10.1097/IAE.0000000000003385. PMID 34934034
- [Derived] Larsen M, Waldstein SM, Priglinger S, Hykin P, Barnes E, Gekkieva M, Das Gupta A, Wenzel A, Mones J; CRYSTAL Study Group. Sustained Benefits from Ranibizumab for Central Retinal Vein Occlusion with Macular Edema: 24-Month Results of the CRYSTAL Study. Ophthalmol Retina. 2018 Feb;2(2):134-142. doi: 10.1016/j.oret.2017.05.016. Epub 2017 Sep 9. PMID 31047340

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No data were excluded from the Full Analysis Set (FAS )analyses because of protocol deviations.
Period: Overall Study
Arm/Group | Ranibizumab Arm
Started | 357
Completed | 307
Not Completed | 50
Not completed — Physician Decision | 8
Not completed — Protocol Violation | 3
Not completed — Death | 5
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 14
Not completed — Adverse Event | 12

BASELINE CHARACTERISTICS:
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 357
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 229

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) at Month 12 Compared to Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. A positive average change from baseline of BCVA indicates improvement
Time Frame: Baseline to month 12
Population: The Full analysis set (FAS) with use of Last Observation Carried Forward (LOCF) consisted of all patients who received at least 1 administration of study treatment and had at least 1 post-baseline assessment for BCVA in the study eye. One patient was excluded from the FAS for not having ≥ 1 post-baseline study eye VA assessment.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 356
Letters | 12.3 (16.72)

2. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) at Month 24 Compared to Baseline
Description: as for outcome 1
Time Frame: Baseline to Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 356
Letters | 12.1 (18.60)

3. Secondary Outcome: Mean Average Change in Best Corrected Visual Acuity (BCVA From Baseline Month 12 and Month 24
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. Mean Average Change: for each patient, first average change is calculated as the average of the changes from baseline to Month 1 over Month 12 (or Month 24). Then, mean average change is calculated as the average of average changes across all patients.
Time Frame: Baseline and Month 1 to 12 or Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 356
letters
  Month 12 | 11.8 (12.44)
  Month 24 | 12.1 (14.20)

4. Secondary Outcome: Mean Average Change in BCVA From First Treatment Interruption (Due to BCVA Stabilization) to Month 12 and Month 24
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. Stability in visual acuity after treatment interruption indicates longer duration of the drug efficacy
Time Frame: Month 12 and Month 24
Population: Full analysis set with use of LOCF consisted of all patients who received at least 1 administration of study treatment and had at least 1 post-baseline assessment for BCVA in the study eye. The number of patients shown was with a value at treatment interruption and an average for the post treatment interruption visits.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 356
Letters
  Month 12 (n=310) | -2.7 (8.04)
  Month 24 (n=331) | -2.5 (8.95)

5. Secondary Outcome: Number of Patients With a BCVA Improvement of ≥1, ≥5, ≥10, ≥15, and ≥30 Letters From Baseline to Month 12 and Month 24 in the Study Eye
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the number of participants who had improvement of ≥1, ≥5, ≥10, ≥15, and ≥30 letters of visual acuity at month 12 as compared with baseline
Time Frame: Month 12 and Month 24
Population: The Full analysis set (FAS) with use of Last Observation Carried Forward (LOCF) consisted of all patients who received at least 1 administration of study treatment and had at least 1 post-baseline assessment for BCVA in the study eye. No data were excluded from the FAS analyses because of protocol deviations.
Measure: Number; unit: Letters
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 356
Letters
  BCVA improvement of >= 1 (Month 12) | 296
  BCVA improvement of >= 5 (Month 12) | 275
  BCVA improvement of >= 10 (Month 12) | 227
  BCVA improvement of >= 15 (Month 12) | 175
  BCVA improvement of >= 30 (Month 12) | 32
  BCVA improvement of >= 1 (Month 24) | 290
  BCVA improvement of >= 5 (Month 24) | 265
  BCVA improvement of >= 10 (Month 24) | 224
  BCVA improvement of >= 15 (Month 24) | 175
  BCVA improvement of >= 30 (Month 24) | 44

6. Secondary Outcome: Number of Patients With a BCVA Value of ≥ 73 Letters (Approximate 20/40 Snellen Chart Equivalent) at Month 12 and Month 24
Description: Best Corrected Visual Acuity (BCVA) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart at baseline and month 12 while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. BCVA above 73 letters at month 12 and month 24 indicates a positive outcome.
Time Frame: Month 12 and Month 24
Population: as for outcome 5
Measure: Number; unit: Letters
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 356
Letters
  Month 12 | 169
  Month 24 | 161

7. Secondary Outcome: Mean Change in Central Reading Center (CRC)-Assessed Central Subfield Thickness (CSFT) From Month 12 and Month 24 Compared to Baseline
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT). The images were reviewed by a central reading center to ensure a standardized evaluation
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 347
Microns
  Change from Baseline at Month 12 | -335.7 (285.02)
  Change from Baseline at Month 24 | -349.1 (275.35)

8. Secondary Outcome: Mean Change in Patient-reported Outcomes in NEI-VFQ-25 Composite and Subscale Scores at Month 12 and Month 24 Compared to Baseline
Description: The survey consists of 25 items representing 11 vision related constructs (general vision, ocular pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision, peripheral vision) plus a single-item general health rating question. The score of each individual question ranges from 0 (worst) to 100 which indicates the best possible response. The composite score and score of each of each construct also range from 0 to 100 as they are calculated as total scores divided by the number of questions. The higher the values of total scores represent better outcome. Scores per visit and of the change descriptively by visit.
Time Frame: Month 12 and Month 24
Population: The Full analysis set (FAS) with use of Last Observation Carried Forward (LOCF) consisted of all patients who received at least 1 administration of study treatment and had at least 1 post-baseline assessment for BCVA in the study eye. The number of patients shown was with a value for both baseline and the post-baseline visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ranibizumab Arm
Number analyzed (Participants) | 350
Score on a scale
  Change from baseline at Month 12 | 6.9 (12.65)
  Change from baseline at Month 24 | 6.6 (14.03)

ADVERSE EVENTS:
Groups:
- Ranibizumab 0.5mg: Intravitreal injection with standard dose of 0.5 mg/0.05mL PRN
Arm/Group | Ranibizumab 0.5mg
Serious Adverse Events (participants affected / at risk) | 64/357
Other Adverse Events (participants affected / at risk) | 244/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg (N=357)
Anaemia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 3
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 3
Cardiopulmonary failure (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 3
Right ventricular failure (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Fellow untreated eye) (Eye disorders) | 1
Cataract (Study eye) (Eye disorders) | 1
Glaucoma (Fellow untreated eye) (Eye disorders) | 1
Glaucoma (Study eye) (Eye disorders) | 2
Hyphaema (Fellow untreated eye) (Eye disorders) | 1
Hyphaema (Study eye) (Eye disorders) | 1
Myopia (Study eye) (Eye disorders) | 1
Retinal haemorrhage (Study eye) (Eye disorders) | 1
Retinal ischaemia (Study eye) (Eye disorders) | 2
Retinal vascular thrombosis (Study eye) (Eye disorders) | 1
Visual acuity reduced (Study eye) (Eye disorders) | 2
Vitreous haemorrhage (Fellow untreated eye) (Eye disorders) | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Death (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Febrile infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Ophthalmic herpes zoster (Fellow untreated eye) (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Intraocular pressure increased (Study eye) (Investigations) | 1
Visual acuity tests abnormal (Study eye) (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain hypoxia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Renal mass (Renal and urinary disorders) | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Aneurysm ruptured (Vascular disorders) | 1
Angiopathy (Vascular disorders) | 1
Diabetic vascular disorder (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg (N=357)
Blepharitis (Study eye) (Eye disorders) | 12
Cataract (Fellow untreated eye) (Eye disorders) | 11
Cataract (Study eye) (Eye disorders) | 15
Conjunctival haemorrhage (Study eye) (Eye disorders) | 24
Dry eye (Fellow untreated eye) (Eye disorders) | 19
Dry eye (Study eye) (Eye disorders) | 22
Eye pain (Study eye) (Eye disorders) | 25
Eyelid oedema (Study eye) (Eye disorders) | 9
Glaucoma (Fellow untreated eye) (Eye disorders) | 10
Glaucoma (Study eye) (Eye disorders) | 11
Macular fibrosis (Study eye) (Eye disorders) | 15
Macular oedema (Study eye) (Eye disorders) | 19
Ocular discomfort (Study eye) (Eye disorders) | 10
Ocular hyperaemia (Study eye) (Eye disorders) | 9
Ocular hypertension (Fellow untreated eye) (Eye disorders) | 8
Ocular hypertension (Study eye) (Eye disorders) | 26
Vision blurred (Study eye) (Eye disorders) | 18
Visual acuity reduced (Study eye) (Eye disorders) | 21
Vitreous detachment (Study eye) (Eye disorders) | 12
Vitreous floaters (Study eye) (Eye disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 11
Injection site pain (Study eye) (General disorders) | 11
Bronchitis (Infections and infestations) | 15
Conjunctivitis (Fellow untreated eye) (Infections and infestations) | 8
Conjunctivitis (Study eye) (Infections and infestations) | 10
Influenza (Infections and infestations) | 17
Lower respiratory tract infection (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 39
Pneumonia (Infections and infestations) | 8
Sinusitis (Infections and infestations) | 9
Tooth infection (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 9
Fall (Injury, poisoning and procedural complications) | 15
Intraocular pressure increased (Fellow untreated eye) (Investigations) | 11
Intraocular pressure increased (Study eye) (Investigations) | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 13
Dizziness (Nervous system disorders) | 11
Headache (Nervous system disorders) | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Hypertension (Vascular disorders) | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety